CLINICAL TRIAL: NCT03765255
Title: Personal Responsibility Education Program Innovative Strategies: Digital Initiative for Youth; An Innovative Youth-Centered Initiative to Improve the Sexual Health and Socio-Economic Well-Being of Youth in Fresno County, California
Brief Title: Personal Responsibility Education Program Innovative Strategies: Digital Initiative for Youth
Acronym: PREIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Youth+Tech+Health (Unknown); Fresno Economic Opportunities Commission (Unknown); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 90AP2688
Record Dates: First submitted 2018-11-13; First posted 2018-12-05 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Reproductive Health; Contraception; Sexually Transmitted Diseases
Keywords: youth; adolescent
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Adolescents will be randomly assigned to treatment or control by cohort (groups of 5-25 adolescents). Adolescents will consent to participation and complete baseline survey prior to randomization. Enrollment will continue by cohort for approximately 2 years. Approximately 15 sites will participate with 2-4 cohorts per site per year.
Who Masked: Outcomes Assessor
Masking Description: The adolescents and the staff enrolling the participants will not know of study assignment until after completing recruitment, consent, and baseline. At that point, they will open an envelope stating if it is a control or treatment cohort. The researcher conducting the outcomes analysis will not know enrollment status of an individual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In the Know (ITK): sexual health education (Experimental): Cohorts/participants in the experimental (treatment) arm receive an intervention that combines 6 hours of in-person sexual health and adolescent development education with an app that includes a resource locator, text message reminders (for one month), goal setting, and other resources.
  Interventions: Other: In the Know: sexual health education
- Control: do not receive ITK intervention (No Intervention): Cohorts/participants in the no intervention arm do not receive either the in-person education or the app. However, after completing the 10 month survey, they will have access to the app and will be invited to participate in the in-person program after the study implementation phase is completed (years 4 and 5).

INTERVENTIONS:
Other: In the Know: sexual health education — The in-person sessions include modules on: sexual and reproductive health (2 hours - anatomy, gender and sexual orientation, pregnancy, contraception, sexually transmitted infections); healthy relationships and life skills (2 hours - communication and negotiation, consent, violence, online dating, goal setting, strengths); and educational and career success (2 hours - educational and career options, applying for scholarships and financial aid, job readiness, resume preparation, interview skills). The app includes: online referrals, personal life plans/goal setting, text message reminders, quizzes, and other resources.
  Arms: In the Know (ITK): sexual health education

SUMMARY:
This randomized control trial (RCT) will assess an innovative demonstration project to improve adolescent sexual and reproductive health among highly mobile and marginalized youth in Fresno County, California. The Digital Initiative for Youth intervention combines existing, in-person, group-based, comprehensive sexual health education with wraparound digital technologies. The technological component was designed by Youth+Tech+Health using a "youth-centered" design approach and the intervention is implemented by Fresno Economic Opportunities Commission (Fresno EOC). The University of California, San Francisco is the external evaluator. The RCT will assess health and behavioral outcomes at three time points (baseline, 4 months, 10 months).

DETAILED DESCRIPTION:
The Digital Initiative for Youth (DIY) is an innovative, youth-centered, digital intervention that aims to improve the health and well-being of adolescents ages 13-19 in Fresno County, California. In particular, it will address the needs of homeless and unstably housed youth, youth of color, sexual minority youth, and Native American youth using a trauma-informed approach and positive youth development framework.

DIY combines existing, in-person, group-based, comprehensive sexual health education with an app designed in consultation with youth. DIY is built on three strategies: positive youth development, youth-centered design, and wraparound technologies. It will focus on four main areas: sexual health and contraceptive use, healthy relationships, educational and career development, and life skills. The intervention includes six hours of in-person education and an app that includes a resource locator, goal setting, text message reminders, and additional information and referrals.

This study is funded through the Personal Responsibility Education Program Innovative Strategies (PREIS), which is administered by the Family and Youth Services Bureau, part of Health and Human Services,

Fresno EOC is responsible for site and participant recruitment as well as the implementation of the intervention. Participants are randomized at the cohort (group) level. All control group participants will be invited to participate after completion of the long-term follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Speak/understand Spanish or English
* Live within Fresno County, California at baseline (may move out afterward)
* Age between 13-19
* Have access to a smart phone or internet (does not need to own)

Exclusion Criteria:

* Do not live in Fresno County, California at baseline
* Do not speak or understand Spanish or English
* Severe mental health issues that prevent them from participating

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1260 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Self-reported condom/contraceptive use or no sex in the last three months on survey | Short term follow up (3 months)
  Answered some or all of the time to: In the past 3 months, how often did you or a partner use birth control when you had vaginal sex OR In the past 3 months, how often did you use condoms when you had anal sex? Respondents complete computer-based survey. Survey developed by University of California, San Francisco (UCSF).
Self-reported use of any clinic services in the last three months on survey | Long-term follow up (9 months)
  Checked any services from survey list after question, "Please check all of the services you have received from a doctor, counselor, therapist, social worker, or clinic in the past 3 months." Respondents complete computer-based survey. Survey developed by UCSF.

SECONDARY OUTCOMES:
Self-reported sexual risk behavior on survey | Short-term follow up (3 months)
  Respondents provide number of sexual partners in past 3 months on computer-based survey. Survey developed by UCSF.
Self-reported knowledge of local clinical services on survey | Short-term follow up (3 months)
  Answered yes to question on computer-based survey: "Have you heard of a clinic or doctor in your community where teens can get sexual health information and services such as condoms, birth control, pregnancy tests, sexually transmitted infection (STI) tests/treatment, and/or HIV tests?" Survey developed by UCSF.

OTHER OUTCOMES:
Self-reported healthy relationship skills on survey | Short-term follow up (3 months)
  Increased number of correct answers on knowledge about healthy relationships questions on computer-based survey between baseline and short-term follow up. Survey developed by UCSF.
Self-reported career and education skills on survey | Long-term follow up (9 months)
  Respondents answer they are or have been enrolled in career training, internships, or educational support. Respondents complete computer-based survey. Survey developed by UCSF.
Self-reported goal setting skills on survey | Short-term follow up (3 months)
  Aggregate responses to "worked on an educational and/or career goal" and "made plans to reach your goals" on computer-based survey. Survey developed by UCSF.

CONTACTS AND LOCATIONS:
Overall Officials: Mara J Decker, DrPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Fresno Economic Opportunities Commission, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We are in discussion with our federal sponsor to determine the sharing plan for a public use dataset.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available on or before October 2021.
Access Criteria: Requirements for access is being developed by the federal sponsors.

DOCUMENTS (1):
  • Informed Consent Form (2017-09-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT03765255/ICF_000.pdf